CLINICAL TRIAL: NCT01613209
Title: Sevicontrol-1: Efficacy and Safety of a Fixed Combination of Olmesartan 40 mg / Amlodipine 10 mg in Patients With Insufficiently Controlled Hypertension Under Monotherapy With Candesartan 32 mg - an Open Phase IIIb Trial
Brief Title: Sevicontrol-1: Efficacy and Safety of a Fixed Combination of Olmesartan/ Amlodipine
Acronym: Sevicontrol1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sevicontrol-1
Record Dates: First submitted 2012-05-30; First posted 2012-06-07 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension
Keywords: Hypertension; ABPM; office blood pressure; olmesartan; amlodipine; fixed combination; time of intake
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; olmesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olmesartan/Amlodipin fixed combination (Experimental)
  Interventions: Drug: Candesartan cilexetil; Drug: Olmesartan/Amlodipin

INTERVENTIONS:
Drug: Candesartan cilexetil — candesartan 16 mg tablets p. o. for 14 days (morning), then candesartan 32 mg tablets for 28 day (morning)s,
Drug: Olmesartan/Amlodipin — olmesartan/amlodipine 40/5 mg tablets for 14 days (morning), then olmesartan/amlodipine 40/10 mg tablets for 28 days (morning), then olmesartan/amlodipine 40/10 mg tablets for 42 days (evening)
  Other Names: Sevikar(r)

SUMMARY:
The investigators want to find out whether a recently introduced combination of two blood pressure lowering agents (olmesartan and amlodipine) has a different blood pressure lowering effect than a single active substance. In addition the investigators want to find out whether there is a difference in the changes in blood pressure over the course of a day depending on the time when the medications are taken (in the morning or at night). Male and female patients over 18 years of age may participate.

DETAILED DESCRIPTION:
Investigation of changes in blood pressure after six weeks therapy with a fixed combination of 40 mg olmesartan and 10 mg amlodipine compared to a monotherapy with 32 mg candesartan. Investigation of changes in dipping-profile after a further six weeks of therapy with the fixed combination when time of intake is switched from morning to evening.

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension, i. e. systolic OPM >=140 mmHg at screening and >=160 mmHg after two weeks wash-out

Exclusion Criteria:

* systolic office bp > 180 mm Hg at screening visit

  * known hypertensive retinopathy GIII or IV
  * recent (< 4 weeks ago) myocardial infarction or indication for coronary or peripheral revascularisation
  * type I diabetes or poorly controlled (HbA1c >= 8) type II diabetes
  * chronic heart failure NYHA III or IV
  * prior stroke or TIA
  * creatinine clearance < 60 ml/min or condition after kidney transplant
  * moderately or severely impaired liver function (ALT or AST or bilirubin more than double normal value)
  * women of childbearing potential without highly effective contraception, pregnant or breastfeeding women
  * concomitant therapy with lithium
  * hemodynamically relevant mitral or aortic valve stenosis (>= II°) or hypertrophic obstructive cardiomyopathy
  * concomitant therapy with strong CYP3A4 inhibitors or inductors
  * african patients
  * concomitant severe psychiatric condition that might impair proper intake of study medication
  * life expectancy < 6 months
  * night shift workers
  * known other mandatory indication for treatment with antihypertensive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in ABPM (ambulatory blood pressure measurement) mean daytime systolic values and change in systolic OBPM (office blood pressure measurement). | after six and after 12 weeks
  After 6 weeks therapy with a fixed combination of olmesartan and amlodipine compared to monotherapy with candesartan
change in systolic OBPM | after 6 and after 12 weeks
  After 6 weeks therapy with a fixed combination of olmesartan and amlodipine compared to monotherapy with candesartan: change in systolic OPM.

SECONDARY OUTCOMES:
change in diastolic OBPM | after six and after 12 weeks
  After 6 weeks therapy with a fixed combination of olmesartan and amlodipine compared to monotherapy with candesartan
Change in systolic and diastolic ABPM night mean values | after 6 weeks therapy with fixed combination of olmesartan and amlodipine
  first ABPM to be performed after 2 weeks wash-out followed by six weeks monotherapy with candesartan. Second ABPM to be performed after six weeks therapy with the fixed combination, given in the morning.
change in 24 hr mean values and diastolic day mean value | after six and after 12 weeks
Distribution of patients over the four dipper types | after six and after 12 weeks
Number of patients achieving target values for OBPM and ABPM | after six and after 12 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From screening visit to end of follow-up, up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Lueders, Dr.med., Principal Investigator — Krankenhaus St.-Josef-Stift, Krankenhausstraße 13, D-49661 Cloppenburg
Locations (12):
- Germany (12):
  - Praxis Dr. Loddo, Rastede, Lower Saxony
  - Praxis Dr. Paschmionka, Leipzig, Saxony
  - Praxis Dr. Reimer, Anderbeck
  - Praxis Dr. Heinz, Bergisch Gladbach
  - Praxis Dr. Zemmrich, Berlin
  - Praxis Dr. Biedermann, Blankenhain
  - St.-Josefs-Hospital, Cloppenburg
  - Praxis Dr. Pohl, Dresden
  - Praxis Koßler-Wiesweg, Essen
  - Praxis Dr. Rövenich, Frankfurt
  - Praxis Dr. Strzata, Kapellendorf
  - Praxis Dr. Pitule, Ludwigshafen

IPD SHARING:
Plan to Share IPD: No